CLINICAL TRIAL: NCT04329403
Title: Randomized, Double Blind, Placebo Controlled, Parallel Group Design, Three Arm, Multicentric Study to Evaluate the Efficacy and Safety of Topical Adapalene Gel, 0.1 % in Healthy Males and Nonpregnant Female Subjects With Acne Vulgaris
Brief Title: Clinical Endpoint Bioequivalence Study of Adapalene Gel 0.1%
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Market reasons
Sponsor: Aurobindo Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR191-18
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Test Group (Experimental): Adapalene Gel, 0.1%, applied as thin film once daily for 12 weeks
  Interventions: Drug: Adapalene 0.1% Gel
- Reference Group (Active Comparator): Differin® (Adapalene) Gel, 0.1%, applied as thin film once daily for 12 weeks
  Interventions: Drug: Differin 0.1% Topical Gel
- Placebo Group (Placebo Comparator): Placebo Gel, 0.1%, applied as thin film once daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Adapalene 0.1% Gel — A thin film of the assigned medication to be applied once daily in the evening for 12 weeks
  Arms: Test Group
Drug: Differin 0.1% Topical Gel — A thin film of the assigned medication to be applied once daily in the evening for 12 weeks
  Arms: Reference Group
Other: Placebo — A thin film of the assigned medication to be applied once daily in the evening for 12 weeks
  Arms: Placebo Group

SUMMARY:
To evaluate the therapeutic equivalence of topical Adapalene Gel, 0.1 % and Differin®(Adapalene) Gel, 0.1 % in the treatment of acne vulgaris and to demonstrate the superiority of the efficacy of the test and reference products over the placebo.

DETAILED DESCRIPTION:
Bio-Equivalence study with a clinical endpoint in the treatment of acne vulgaris comparing adapalene cream, 0.1% test product versus the reference listed drug (RLD) and placebo (vehicle) control, each administered as one application once a day in the evening for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant, nonlactating female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris
2. On the face, ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 20 inflammatory lesions (i.e., papules and pustules) AND ≤ 2 nodulocystic lesions (i.e., nodules and cysts)
3. Investigator's Global Assessment (IGA) of acne severity Grade 2, 3, or 4
4. Willing to refrain from use of all other topical acne medications or antibiotics during the 12-week treatment period
5. If female of childbearing potential, willing to use an acceptable form of birth control during the study

Exclusion Criteria:

1. Pregnant, breast feeding or planning a pregnancy
2. Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis)
3. Excessive facial hair (e.g., beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris
4. History of hypersensitivity or allergy to adapalene, retinoids and/or any of the study medication ingredients
5. Use within 6 months prior to baseline or during the study of oral retinoids (e.g., Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed)
6. Use for less than 3 months prior to baseline of estrogens or oral contraceptives; use of such therapy must remain constant throughout the study
7. Use on the face within 1 month prior to baseline or during the study of 1) cryo destruction or chemo destruction, 2) dermabrasion, 3) photodynamic therapy, 4) acne surgery, 5) intralesional steroids, or 6) x-ray therapy
8. Use within 1 month prior to baseline or during the study of 1) systemic steroids, 2) systemic antibiotics, 3) systemic treatment for acne vulgaris (other than oral retinoids, which require a 6-month washout), or 4) systemic anti-inflammatory agents
9. Use within 2 weeks prior to baseline or during the study of 1) topical steroids, 2) topical retinoids, 3) topical acne treatments including over-the-counter preparations, 4) topical anti-inflammatory agents, or 5) topical antibiotics

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Mean percent change from baseline in the inflammatory lesion count. | 12 weeks
  Mean percent change compared to baseline inflammatory lesion count (papules and pustules) at Day 84 in per protocol population.
Mean percent change from baseline in the non-inflammatory lesion count. | 12 weeks
  Mean percent change compared to baseline non-inflammatory lesion count (open and closed comedones) at Day 84 in per protocol population.

SECONDARY OUTCOMES:
Proportion of subjects with a clinical response as success or failure | 12 weeks
  Success will be defined as IGA score that is at least 2 grades less than the baseline assessment. Failure is defined as an IGA score that is the same, higher or one grade lower than the baseline assessment.
Change in lesion count | 12 weeks
  Percentage of subjects who achieved at least 50 % reduction in lesion counts (inflammatory, non-inflammatory and total lesion count)